CLINICAL TRIAL: NCT05089734
Title: Open-Label, Global, Multicenter, Randomized, Phase 3 Study of Sacituzumab Govitecan Versus Docetaxel in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) With Progression on or After Platinum-Based Chemotherapy and Anti-PD-1/PD-L1 Immunotherapy
Brief Title: Study of Sacituzumab Govitecan (SG) Versus Docetaxel in Participants With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Acronym: EVOKE-01
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-577-6153; jRCT2051220119 (Registry Identifier: Japan Registry of Clinical Trials); 2024-512148-50 (Other: European Medicines Agency)
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sacituzumab govitecan; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab Govitecan-hziy (SG) (Experimental): Participants will receive SG 10 mg/kg on Days 1 and 8 of a 21-day cycle (ie, 2 weekly doses plus 1 week without treatment) until progressive disease (PD), death, unacceptable toxicity, or another treatment discontinuation criterion is met.
  Interventions: Biological: Sacituzumab Govitecan-hziy (SG)
- Docetaxel (Active Comparator): Participants will receive docetaxel 75 mg/m^2 on Day 1 of a 21-day cycle (ie, once every 3 weeks) until PD, death, unacceptable toxicity, or another treatment discontinuation criterion is met.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: Sacituzumab Govitecan-hziy (SG) — Administered intravenously
  Other Names: IMMU-132; GS-0132
  Arms: Sacituzumab Govitecan-hziy (SG)
Drug: Docetaxel — Administered intravenously
  Arms: Docetaxel

SUMMARY:
The goal of this clinical study is to compare the study drug, sacituzumab govitecan-hziy (SG), versus docetaxel in participants with advanced or metastatic (cancer that has spread) non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Key Inclusion Criteria:

* Pathologically documented non-small cell lung cancer (NSCLC) with documented evidence of Stage 4 NSCLC disease at the time of enrollment (based on the American Joint Committee on Cancer, Eighth Edition).
* Epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), and programmed death protein 1 (PD-1)/programmed death ligand 1 (PD-L1) results are required. Testing prior to enrollment. Resulting for other actionable genomic alterations is recommended and to be performed as per local standard of care and availability of targeted treatment. For patients with squamous cell carcinoma, EGFR and ALK testing is optional.
* Must have progressed after platinum-based chemotherapy in combination with anti-PD-1/PD-L1 antibody OR platinum-based chemotherapy and anti-PD-1/PD-L1 antibody (in either order) sequentially.

  * No additional treatments are allowed in the recurrent/metastatic setting for individuals with no actionable genomic alterations.
  * Individuals with EGFR, ALK, or any other known actionable genomic alterations must have also received treatment with at least 1 locally approved and available tyrosine kinase inhibitor 1(TKI) appropriate to the genomic alteration.
  * Documented radiographic disease progression while on or after receiving the most recent treatment regimen for advanced or metastatic NSCLC.
* Measurable disease based on computed tomography (CT) or magnetic resonance imaging (MRI) as assessed by the investigator in accordance with per RECIST Version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 before randomization.
* Adequate hematologic counts without transfusional or growth factor support within 2 weeks of study drug initiation (hemoglobin ≥ 9 g/dL, absolute neutrophil count ≥ 1500/mm^3, and platelets ≥ 100,000/μL).
* Adequate hepatic function (bilirubin ≤ 1.5 x upper limit of normal (ULN), aspartate aminotransferase and alanine aminotransferase ≤ 2.5 ULN or ≤ 5 x ULN if known liver metastases, and serum albumin > 3 g/dL).
* Creatinine clearance of at least 30 mL/min as assessed by the Cockcroft-Gault equation.
* Male individuals and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.

Key Exclusion Criteria:

* Mixed small-cell lung cancer and NSCLC histology.
* Positive serum pregnancy test or women who are lactating.
* Received a prior anticancer biologic agent within 4 weeks prior to enrollment or have received prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to enrollment and have not recovered (ie, > Grade 2 is considered not recovered) from adverse events (AEs) at the time of study entry. Individuals participating in observational studies are eligible.
* Have not recovered (ie, > Grade 2 is considered not recovered) from AEs due to a previously administered agent.
* Previously received treatment with any of the following:

  * Topoisomerase 1 inhibitors. Any agent including an antibody-drug conjugate (ADC) containing a chemotherapeutic agent targeting topoisomerase 1
  * Trop-2-targeted therapy
  * Docetaxel as monotherapy or in combination with other agents
* Active second malignancy
* NSCLC that is eligible for definitive local therapy alone.
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (ie, pulmonary emboli within 3 months of enrollment, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc); any autoimmune, connective tissue, or inflammatory disorders with pulmonary involvement (ie, rheumatoid arthritis, Sjogren syndrome, sarcoidosis, etc); or prior pneumonectomy.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Active cardiac disease
* Active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or gastrointestinal perforation within 6 months of enrollment.
* Active serious infection requiring antibiotics.
* Positive HIV-1 or HIV-2 antibody with detectable viral load OR taking medications that may interfere with SN-38 metabolism.
* Positive for hepatitis B surface antigen. Individuals who test positive for hepatitis B core antibody will require hepatitis B virus DNA by quantitative polymerase chain reaction for confirmation of active disease.
* Positive hepatitis C antibody and detectable hepatitis C viral load.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (227):
- United States (37):
  - Alaska Oncology and Hematology, LLC., Anchorage, Alaska
  - USOR - Arizona Oncology Associates Tucson - Wilmot, Tucson, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Florida Cancer Specialists (Administration and Drug Shipment), Fort Myers, Florida
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Siouxland Regional Cancer Center dba June E. Nylen Cancer Center, Sioux City, Iowa
  - Kansas City VA Medical Center, Westwood, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Maryland Oncology Hematology, P.A., Clinton, Maryland
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Park Nicollet Frauenshuh Cancer Center, Saint Paul, Minnesota
  - Nebraska Hematology - Oncology, Lincoln, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Broome Oncology, LLC, Johnson City, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - W.G (Bill) Hefner VAMC, Salisbury, North Carolina
  - Zangmeister Cancer Center, Columbus, Ohio
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology - Denison, Denison, Texas
  - Texas Oncology - Denton South, Denton, Texas
  - Texas Oncology Cancer Care and Research Center, McAllen, Texas
  - USOR - Texas Oncology - McKinney, McKinney, Texas
  - Texas Oncology - Paris, Paris, Texas
  - Texas Oncology-Plano East, Plano, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - Shenandoah Oncology Associates, PC, Winchester, Virginia
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (12):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Southern Highlands Cancer Centre, Bowral, New South Wales
  - St Vincent's Public Hospital, Darlinghurst, New South Wales
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Gallipoli Medical Research Foundation, Greenslopes, Queensland
  - Flinders Medical centre, Bedford Park, South Australia
  - Icon Cancer Centre, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Joondalup Health Campus, Joondalup, Western Australia
  - ir Charles Gairdner Hospital, Perth, Western Australia
- Austria (4):
  - Medizinische Universität Innsbruck, Medizinische Universitat Innsbruck, Universitatsklinik fur Innere Medizin V, Hamatologie und Onkolgie, Innsbruck
  - Muellner Hauptstrabe 48, Salzburg
  - zuniklinikum Salzburg, Landeskrankenhaus, Universitatsklinik fur Innere Medizin III der PMU, Salzburg
  - Klinik Floridsdorf, Karl Landsteiner Institute fur Lungenforschung und Pneumologische onkologie (LFPO) Abteilung Fur Innere Medizin un Pneumologie, Vienna
- Belgium (6):
  - Algemeen Ziekenhuis Klina, Brasschaat
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Algemeen Ziekenhuis Sint-Lucas, Ghent
  - Az Maria Middelares Ghent, Ghent
  - CHU Ambroise Pare, Mons
- Brazil (9):
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí
  - Catatina Pesquisa Clinica - Clinica de Neoplasias Litoral, Itajaí
  - Centro de Pesquisas Clinicas da Fundacao Doutor Amaral Carvalho, Jaú
  - Hospital de Clínicas de Porto Alegre - HCPA, Porto Alegre
  - Centro Gaucho Integrado de Oncologia, Hematologia, Ensino e Pesquisa, Porto Alegre
  - Nucleo de Pesquisa da Rede Sao Camilo-Instituto Brasileiro de controle do cancer-IBC, São Paulo
  - A Beneficência Portuguesa de São Paulo, São Paulo
  - Instituto do Câncer do Estado de São Paulo "Octavio Frias de Oliveira" - ICESP, São Paulo
- Canada (5):
  - Royal Victoria Regional Health Centre, Barrie
  - William Osler Health System-Brampton Civic Hospital, Brampton
  - McGill University Health Centre, Montreal
  - Required Centre Hospitalier Regional de Rimouski, Rimouski
  - Windsor Regional Hospital Cancer Program, Windsor
- France (24):
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - APHP-Hopital Ambroise-Pare, Boulogne-Billancourt
  - CHU de CAEN, Caen
  - Centre Francois Baclesse, Calvados
  - Centre Hospitalier de Chauny, Chauny
  - CHU-Hopital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Centre Hospitalier Annecy Genevois, Epagny Metz-tessy
  - Centre Hospitalier Departemental Vendee, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - CHU de Lille, Lille
  - Hopital Dupuytren (CHU de Limoges), Limoges
  - Chu Montpellier Hopital Arnaud de Villeneuve, Montpellier
  - GHR Sud Alsace - Hopital Emile Muller, Mulhouse
  - Institut Curie, Paris
  - CHU de Bordeaux Hopital Haut leveque, Pessac
  - Hospices Civils de Lyon, Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Rouen - Hopitel Charles Nicolle, Rouen
  - Institut de Cancérologie de l'Ouest - Paysde Loire (site SAINT HERBLAIN), Saint-Herblain
  - Hopital Foch, Saint-Herblain
  - Institut Cancérologie Strasbourg Europe, Strasbourg
  - CHITS-Hopital Sainte Musse, Toulon
- Germany (11):
  - Stadtisches Klinikum Braunschweig gGmbH Medizinische Klinik III Hamatologie und Onkologie, Braunschweig
  - Klinikum Esslingen GmbH Klinik fur Kardiologie,Angiologie und Pneumologie, Esslingen am Neckar
  - Asklepios Klinikum Harburg, Thoraxzentrum Hamburg - Lungenabteilung, Hamburg
  - Studiengeselischaft Hamato-Onkologie Hamburg, Hamburg
  - Onkologische Schwerpunktpraxis Heilbronn, Heilbronn
  - Lungenfachklink Immenhausen, Immenhausen
  - Klinikum Kassel Klinik Für Hämatologie Onkologie Und Immunologie, Kassel
  - Universitatsklinikum Schleswig-Holstein - Campus Lubeck, Medizinische Klinik III (Studienzentrum Pneumologie), Lübeck
  - University Hospital Mannheim, Department of Personalized Medical Oncology with Section Thoracic Oncology, Mannheim
  - Asklepios-Fachkliniken Munchen-Gauting, Zentrum fur Pneumologie und Thoraxchirurgie, Munchen-Gauting
  - Sana Klinikum Offenbach, Medizinische Klinik IV fur Hamatologie und internistische Onkologie, Offenbach
- Greece (8):
  - Henry Dunant Hospital Center, 4th Oncology Department, Athens
  - General Hospital of Chest Diseases "I Sotiria", 3rd Internal Medicine Department of Athens University - Oncology Unit, Athens
  - Metropolitan General, Oncology department, Cholargós
  - General Oncology Hospital of Kifisia "Agioi Anargyroi", 2nd Department of Medical Oncology, Heraklion
  - University General Hospital of Larissa, Oncology Department-1St Internal Medical Division, Larissa
  - General Oncology Hospital of Kifisia "Agioi Anargyroi", 2nd Department of Medical Oncology, Nea Kifissia
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki
- Israel (6):
  - Samson Assuta Ashdod University Hospital, Ashdod
  - Soroka Medical Center, Beersheba
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Shamir Medical Center (Assaf Harofeh), Tzrifin
- Italy (12):
  - ASST Papa Giovanni XXIII, Oncologia Medica, Bergamo
  - Azienda Socio Sanitaria Territoriale (ASST) degli Spedali Civili di Brescia, Brescia
  - AOU Policlinico G Rodlico-Oncologia Medica, Catania
  - AOU mater Domini, UOC Oncologia Medica e Oncologia Medica Trazionale, Catanzaro
  - ASST Cremona, Cremona
  - Instituto Europeo di Oncologia, Milan
  - ASST Grande Ospedale Metropolitano Niguarda SC Oncologia, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinico Universitario Campus Bio-Medico, UOC Oncologia Medica, Roma
  - UOC Oncologia, San Giovanni Rotondo
  - ASST Bergamo Ovest- ospedale di Treviglio-u.o. Oncologia, Treviglio
  - SC Oncologia -ASST SETTE LAGHI, Varese
- Japan (34):
  - National Hospital Organization Asahikawa Medical Center, Asahikawa
  - National Cancer Center Hospital, Chūō
  - Fukui Prefectural Hospital, Fukui
  - Kansai Medical University Hospital, Hirakata
  - Hiroshima University Hospital, Hiroshima
  - Kobe City Medical Center General Hospital, Hyōgo
  - National Hospital Organization Himeji Medical Center, Hyōgo
  - Nippon Medical School Chiba Hokusoh Hospital, Inzai
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni
  - Kagoshima University Hospital, Kagoshima
  - Kanagawa Prefectural Hospital Organization Kanagawa Cardiovascular and Respiratory Center, Kanagawaken
  - Kanazawa University Hospital, Kanazawa
  - National Cancer Center Hospital East, Kashiwa
  - Saitama Cancer Center, Kitaadachi-gun
  - The Cancer Institute Hospital of JFCR, Kōtō City
  - Kurume University Hospital, Kurume
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Shikoku Cancer Center, Matsuyama
  - Miyagi Cancer Center, Miyagi
  - Nagasaki University Hospital, Nagasaki
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Osakasayama-Shi
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai
  - Centor Hospital of the National Center for Global Health and Medicine, Shinjuku-Ku
  - Shizuoka Cancer Center, Sunto-gun
  - National Hospital Organization Osaka Toneyama Medical Center, Toyonaka
  - Tochigi Cancer Center, Utsunomiya
  - Japanese Red Cross Wakayama Medical Center, Wakayama
  - Yokohama Municipal Citizen's Hospital, Yokohama
  - Kanagawa Cancer Center, Yokohama
  - Tottori University Hospital, Yonago
- Mexico (3):
  - Panamerican Clinical Research S.A. de C.V, Guadalajara
  - Actualidad Basada en la Investigación del Cáncer, Guadalajara
  - Cryptex Investigación Clínica, S.A. de C.V., Mexico City
- Netherlands (5):
  - Amphia Hospital, Breda
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Erasmus MC, Rotterrdam
  - Haaglanden Medical Centre, The Hague
  - Elisabeth-TweeSteden Ziekenhuis (ETZ), Tilburg
- Poland (4):
  - Przychodnia Lekarska Komed Roman Karaszewski, Konin
  - Instytut MSF Sp. z o.o., Lodz
  - Centrum Medyczne Mrukmed, Rzeszáw
  - Marzowiecki Szpital Wojewodzki sw Jana Pawla II Wsiedicach sp. z.o.o Siedickie centrum onkoiogii, Siedlce
- Portugal (7):
  - Instituto Português de Oncologia de Coimbra Francisco Gentil, Coimbra
  - Centro Hospitalar Universitário Lisboa Norte - Hospital Pulido Valente, Lisbon
  - Fundacao Champalimaud, Lisbon
  - Senhora da Hora, Matosinhos Municipality
  - Hospital CUF Porto, Porto
  - Centro Hospitalar Universitario do Porto, Porto
  - Instituto Portugues de Oncologia do Porto, Porto
- Puerto Rico (2):
  - Pan American Center For Oncology Trials, LLC, San Juan, PR
  - Ad-Vance Medical Research, LLC, Ponce
- Spain (22):
  - Complejo Hospitalario Universitario A Coruna. Hospital Teresa Herrera, A Coruña
  - Institut Catala d'Oncologia Badalona, ICO Badalona, Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Institut Catala D'Oncologia (ICO L'Hospitalet) Hospital Duran i Reynals, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Institut Catala d'Oncologia de Girona, Girona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundacion Jimenez Dias, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinical San Carlos, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Hospital universitario la paz, Madrid
  - Hospital Regional Universitario de Malaga-Hospital Civil, Málaga
  - Hospital Clinicl universitario virgen de la Arrixaca, Murcia
  - Clinica Universidad de Navarra-Pamplona, Pamplona
  - Hospital de Sabadell, Sabadell
  - Hospital Virgen de Valme, Seville
  - Hospital universitario Virgen Macarena, Seville
  - Hospital Universitario la Fe, Valencia
- Turkey (Türkiye) (9):
  - Hacettepe Üniversitesi Hastanesi, Ankara
  - Memorial Ankara Hastane, Ankara
  - Acibadem Bursa Hastanesi, Bursa
  - Ankara Sehir Hastanesi, Dikimevi- Ankara
  - Trakya Üniversitesi Sağlık Araştırma ve Uygulama Merkezi, Edirne
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - T.C. Saglik Bakanligi Goztepe Prof. Dr Suleyman Yalcin Sehir Hastanesi, Kadıköy
  - Acibadem Maslak Hastanesi, Sarıyer
  - Gazi Universitesi Gazi Hastanesi, Yenimahalle
- United Kingdom (7):
  - University Hospital Birmingham NHS Trust, Birmingham Heartlands Hospital, Birmingham
  - East Suffolk and North Essex NHS Foundation Trust, Colchester
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - St James University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Barts Health NHS Trust, London
  - The Christie NHS Foundation, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paz-Ares LG, Juan-Vidal O, Mountzios GS, Felip E, Reinmuth N, de Marinis F, Girard N, Patel VM, Takahama T, Owen SP, Reznick DM, Badin FB, Cicin I, Mekan S, Patel R, Zhang E, Karumanchi D, Garassino MC. Sacituzumab Govitecan Versus Docetaxel for Previously Treated Advanced or Metastatic Non-Small Cell Lung Cancer: The Randomized, Open-Label Phase III EVOKE-01 Study. J Clin Oncol. 2024 Aug 20;42(24):2860-2872. doi: 10.1200/JCO.24.00733. Epub 2024 May 31. PMID 38843511
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-577-6153

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe, North America, Brazil, Israel, Japan, Turkey, Australia, and Puerto Rico.
Pre-assignment Details: 784 participants were screened. Data submitted represent interim analysis performed on data collected by the Primary Completion Date. Complete data will be submitted in May 2026.
Groups:
- Sacituzumab Govitecan (SG): Participants received sacituzumab govitecan 10 mg/kg of body weight, administered as a slow intravenous (IV) infusion on Days 1 and 8 of a 21-day treatment cycle until progressive disease (PD), death, unacceptable toxicity, or another treatment discontinuation criterion was met (up to 18.7 months).
- Docetaxel: Participants received docetaxel 75 mg/m^2, administered as IV infusion on Day 1 of a 21-day treatment cycle (ie, once every 3 weeks) until PD, death, unacceptable toxicity, or another treatment discontinuation criterion was met (up to 19.8 months).
Period: Overall Study
Arm/Group | Sacituzumab Govitecan (SG) | Docetaxel
Started | 299 | 304
Completed | 0 | 0
Not Completed | 299 | 304
Not completed — Still on study | 122 | 101
Not completed — Death | 161 | 179
Not completed — Withdrew consent | 11 | 24
Not completed — Lost to Follow-up | 5 | 0

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) Analysis Set included all randomized participants according to the treatment arm to which the participant was randomized.
Groups:
- Sacituzumab Govitecan (SG): Participants received sacituzumab govitecan 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until PD, death, unacceptable toxicity, or another treatment discontinuation criterion was met (up to 18.7 months).
Arm/Group | Sacituzumab Govitecan (SG) | Docetaxel | Total~(N=584)
Number analyzed (Participants) | 299 | 304 | 603
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9.2) | 64 (9.3) | 64 (9.3)
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 65 years | 136 | 161 | 297
  >=65 years | 163 | 143 | 306
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 88 | 193
  Male | 194 | 216 | 410
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Asian | 17 | 26 | 43
  Race: Black | 6 | 7 | 13
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: White | 229 | 216 | 445
  Race: Other | 3 | 4 | 7
  Race: Not Reported | 44 | 49 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 24 | 22 | 46
  Ethnicity: Not Hispanic or Latino | 266 | 268 | 534
  Ethnicity: Not Reported | 9 | 14 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 73 | 66 | 139
  France | 55 | 65 | 120
  United States | 32 | 28 | 60
  Japan | 15 | 22 | 37
  Italy | 20 | 14 | 34
  Germany | 15 | 15 | 30
  Greece | 11 | 15 | 26
  Turkey | 12 | 11 | 23
  Australia | 6 | 14 | 20
  United Kingdom | 8 | 13 | 21
  Canada | 10 | 5 | 15
  Netherlands | 8 | 8 | 16
  Brazil | 7 | 6 | 13
  Belgium | 6 | 8 | 14
  Portugal | 8 | 4 | 12
  Austria | 4 | 4 | 8
  Poland | 4 | 3 | 7
  Israel | 4 | 1 | 5
  Mexico | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization until the date of death from any cause. OS was estimated using Kaplan-Meier estimate. Participants without documentation of death were censored on the date they were last known to be alive.
Time Frame: Up to 24.4 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan (SG) | Docetaxel
Number analyzed (Participants) | 299 | 304
months | 11.1 [9.4 to 12.3] | 9.8 [8.1 to 10.6]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan (SG) vs Docetaxel; Test type: Superiority; p = 0.0534, Log Rank — Stratified log-rank test adjusted for stratification factors: histology and best response to last prior immune therapy received; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.68 to 1.04]

2. Secondary Outcome: Progression-free Survival (PFS) Assessed by Investigator Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS is defined as the time from the date of randomization until the date of objective disease progression (PD) or death from any cause, whichever occurs first as assessed by RECIST v.1.1. As per RECIST 1.1, PD was defined as: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum measured while on study (this included the baseline sum if that was the smallest on study), in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm or the appearance of of 1 or more new lesions or unequivocal progression of existing non-target lesions. Participants who did not have documented disease progression and did not die were censored at their last tumor assessment date. Kaplan-Meier estimate was used for analysis.
Time Frame: Up to 24.4 months
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan (SG) | Docetaxel
Number analyzed (Participants) | 299 | 304
months | 4.1 [3.0 to 4.4] | 3.9 [3.1 to 4.2]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan (SG) vs Docetaxel; Test type: Superiority; p = 0.1938, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.77 to 1.11]

3. Secondary Outcome: Objective Response Rate (ORR) Assessed by Investigator Per RECIST Version 1.1
Description: ORR was defined as the percentage of participants who achieved a complete response (CR) or partial response (PR) that was confirmed at least 4 weeks later as assessed by RECIST v.1.1. As per RECIST 1.1 CR was defined as: Disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal; PR was defined as: At least 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 24.4 months
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sacituzumab Govitecan (SG) | Docetaxel
Number analyzed (Participants) | 299 | 304
percentage of participants | 13.7 [10.0 to 18.1] | 18.1 [13.9 to 22.9]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan (SG) vs Docetaxel; Test type: Superiority; p = 0.9255, Cochran-Mantel-Haenszel — The 1-sided p-value is calculated using Cochran Mantel-Haenszel test adjusted for randomization stratification factors of histology, and best response to last prior immune therapy received; Difference in Proportions = -4.3, 95% CI 2-sided [-10.1 to 1.5]

4. Secondary Outcome: Duration of Response (DOR) Assessed by Investigator Per RECIST Version 1.1
Description: DOR is defined as the time from the first documentation of CR or PR to the earlier of the first documentation of PD or death from any cause (whichever comes first) as assessed by RECIST v. 1.1. As per RECIST 1.1 CR was disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal; PR was at least 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD, and PD was at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum measured while on study (this included the baseline sum if that was the smallest on study), in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm or the appearance of of 1 or more new lesions or unequivocal progression of existing non-target lesions. Kaplan-Meier estimate was used for analysis.
Time Frame: Up to 24.4 months
Population: Participants in the ITT Population who achieved confirmed complete or partial response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan (SG) | Docetaxel
Number analyzed (Participants) | 41 | 55
months | 6.7 [4.4 to 9.8] | 5.8 [4.1 to 8.3]

5. Secondary Outcome: Disease Control Rate (DCR) Assessed by Investigator Per RECIST Version 1.1
Description: DCR was defined as the percentage of participants who achieved a CR, PR,or stable disease(SD)as assessed by RECIST v.1.1. Per RECIST 1.1 CR was disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal;PR was at least 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD,taking as reference the smallest sum LD since the treatment started and persistence of 1 or more nontarget lesion(s).PD was at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum measured while on study (this included the baseline sum if that was the smallest on study),in addition of increase of 20% sum also demonstrate an absolute increase of at least 5 mm or appearance of 1 or more new lesions or unequivocal progression of existing non-target lesions.
Time Frame: Up to 24.4 months
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sacituzumab Govitecan (SG) | Docetaxel
Number analyzed (Participants) | 299 | 304
percentage of participants | 67.6 [61.9 to 72.8] | 67.1 [61.5 to 72.4]

6. Secondary Outcome: Percentage of Participants Who Experienced Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participants administered a medicinal product that does not necessarily have a causal relationship with this treatment. TEAEs were defined as any AEs that begin or worsen on or after the start of study drug through 30 days after the last dose of the study drug. The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 5.0.
Time Frame: Up to 3.5 years
Reporting Status: Not Posted, anticipated posting 2026-05

7. Secondary Outcome: Percentage of Participants Who Experienced Grade 3 or 4 Treatment Emergent Laboratory Abnormalities Post-Baseline
Description: Blood samples were collected for hematology, serum chemistry, and the laboratory abnormalities were assessed. A treatment-emergent laboratory abnormality was defined as an increase of at least 1 toxicity grade from baseline at any time postbaseline up to and including the date of last study drug dose plus 30 days.The most severe graded abnormality observed post-baseline for each graded test was counted for each participant. Safety as assessed by grading of laboratory values and AEs according to the National Cancer Institutes' Common Terminology Criteria for Adverse Events (NCI CTCAE) covering grades 0-5 (0=Normal, 1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening, 5=Death). The percentage of participants with worst postbaseline grades 3 or 4 will be reported.
Time Frame: Up to 3.5 years
Reporting Status: Not Posted, anticipated posting 2026-05

8. Secondary Outcome: Time to First Deterioration in Shortness of Breath Domain as Measured by Non-small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ)
Description: The NSCLC-SAQ is a participant reported outcome with seven items assessing five symptom concepts of NSCLC: cough, pain, dyspnea, fatigue, and appetite. Each item is rated using a five-point verbal rating scale from "No <symptom> At All" to "Very severe <symptom>" or from "Never to Always" depending on the item's question structure relative to either intensity or frequency, corresponding to a score of 0 to 4, with total score ranging from 0 to 20. The dyspnea (shortness of breath) item uses a "Never(0) to Always(4)" rating scale with higher score indicating higher frequency of dyspnea. Time to deterioration (TTD) was defined as the time from date of randomization to the first date a participant achieves 2-point deterioration from baseline. For shortness of breath domain, a 1-point or greater worsening from baseline represents a clinically meaningful deterioration. Kaplan-Meier estimate was used for analysis.
Time Frame: Up to 24.4 months
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan (SG) | Docetaxel
Number analyzed (Participants) | 299 | 304
months | 2.8 [2.2 to 4.0] | 2.1 [1.6 to 2.9]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan (SG) vs Docetaxel; Test type: Superiority; p = 0.0020, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.61 to 0.91]

9. Secondary Outcome: Time to First Deterioration in NSCLC-SAQ Total Score
Description: The NSCLC-SAQ is a participant reported outcome measure with seven items assessing five symptom concepts of NSCLC: cough, pain, dyspnea, fatigue, and appetite. Each item is rated using a five-point verbal rating scale from "No <symptom> At All" to "Very severe <symptom>" or from "Never to Always" depending on the item's question structure relative to either intensity or frequency, corresponding to a score of 0 to 4. A total score sums all five domain scores at each visit. If any domain score was missing, the score was not computed. The total score ranges between 0 and 20, with higher scores indicating more severe symptoms. TTD was defined as the time from date of randomization to the first date a participant achieves 2-point deterioration from baseline. For NSCLC-SAQ total score, a 2-point or greater worsening from baseline represents a clinically meaningful deterioration. Kaplan-Meier estimate was used for analysis.
Time Frame: Up to 24.4 months
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sacituzumab Govitecan (SG) | Docetaxel
Number analyzed (Participants) | 299 | 304
months | 3.1 [2.5 to 3.9] | 2.7 [2.1 to 3.5]
Statistical Analysis 1: Comparison: Sacituzumab Govitecan (SG) vs Docetaxel; Test type: Superiority; p = 0.0125, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.66 to 0.97]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events: Up to 24.4 months
Description: Adverse Events: The Safety Analysis Set included all participants who received at least 1 dose of any study drug, with treatment assignments designated according to the actual treatment received.; All-Cause Mortality: The ITT Analysis Set included all randomized participants according to the treatment arm to which the participant was randomized.
Arm/Group | Sacituzumab Govitecan (SG) | Docetaxel
All-Cause Mortality (participants affected / at risk) | 168/299 | 187/304
Serious Adverse Events (participants affected / at risk) | 137/296 | 124/288
Other Adverse Events (participants affected / at risk) | 283/296 | 267/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan (SG) (N=296) | Docetaxel (N=288)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 20 | 24
Leukopenia (Blood and lymphatic system disorders) | 3 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 10 | 10
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 2
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 14 | 3
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 3 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Chest pain (General disorders) | 1 | 1
Death, not otherwise specified (General disorders) | 1 | 4
Fatigue (General disorders) | 4 | 1
Gait disturbance (General disorders) | 2 | 0
Gait inability (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 6 | 0
Hyperthermia (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 2 | 1
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 5
Vascular stent thrombosis (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 2 | 2
Covid-19 pneumonia (Infections and infestations) | 0 | 3
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 2 | 0
Large intestine infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 1
Pleural infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 13 | 16
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 5
Sepsis (Infections and infestations) | 5 | 1
Septic shock (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
General physical condition abnormal (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Motor dysfunction (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial lung abnormality (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 5
Hypovolaemic shock (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan (SG) (N=296) | Docetaxel (N=288)
Anemia (Blood and lymphatic system disorders) | 119 | 88
Leukopenia (Blood and lymphatic system disorders) | 37 | 62
Lymphopenia (Blood and lymphatic system disorders) | 22 | 31
Neutropenia (Blood and lymphatic system disorders) | 109 | 116
Abdominal pain (Gastrointestinal disorders) | 27 | 14
Constipation (Gastrointestinal disorders) | 86 | 48
Diarrhoea (Gastrointestinal disorders) | 155 | 97
Nausea (Gastrointestinal disorders) | 123 | 75
Stomatitis (Gastrointestinal disorders) | 39 | 57
Vomiting (Gastrointestinal disorders) | 59 | 42
Chest pain (General disorders) | 16 | 12
Fatigue (General disorders) | 167 | 160
Oedema peripheral (General disorders) | 16 | 35
Pyrexia (General disorders) | 35 | 29
Covid-19 (Infections and infestations) | 23 | 18
Pneumonia (Infections and infestations) | 15 | 8
Urinary tract infection (Infections and infestations) | 15 | 8
Alanine aminotransferase increased (Investigations) | 21 | 14
Aspartate aminotransferase increased (Investigations) | 16 | 7
Blood creatinine increased (Investigations) | 16 | 5
Weight decreased (Investigations) | 20 | 11
Decreased appetite (Metabolism and nutrition disorders) | 77 | 69
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 22
Hypokalaemia (Metabolism and nutrition disorders) | 22 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 23 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 15 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 23
Dizziness (Nervous system disorders) | 18 | 17
Dysgeusia (Nervous system disorders) | 14 | 30
Headache (Nervous system disorders) | 25 | 23
Neuropathy peripheral (Nervous system disorders) | 11 | 38
Paraesthesia (Nervous system disorders) | 6 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 46 | 45
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 47
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 18 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 128 | 86
Pruritus (Skin and subcutaneous tissue disorders) | 37 | 11
Rash (Skin and subcutaneous tissue disorders) | 30 | 19
Hypotension (Vascular disorders) | 10 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT05089734/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT05089734/SAP_001.pdf